CLINICAL TRIAL: NCT00997035
Title: The Mycotic Ulcer Treatment Trial II: A Randomized Trial Comparing Oral Voriconazole vs Placebo
Acronym: MUTTII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Hospitals, India (Other); Dartmouth-Hitchcock Medical Center (Other); Lumbini Eye Institute and Research Centre (Other); Bharatpur Eye Hospital (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Thomas M. Lietman, Professor in Residence, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H9332-33965-02_2; U10EY018573 (NIH)
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Corneal Ulcer; Eye Infections, Fungal
Keywords: Fungal Infections; Eye Disease; Fungal Keratitis; Visual Acuity
MeSH Terms: conditions — Corneal Ulcer; Eye Infections, Fungal; Mycoses; Eye Diseases | interventions — Voriconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Voriconazole (Active Comparator)
  Interventions: Drug: Voriconazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Voriconazole — 1% voriconazole (topical) plus 0.01% preservative, 1 drop applied to the affected eye every one hour while awake for 1 week, then every 2 hours while awake until three weeks after enrollment.
  5% natamycin (topical), 1 drop applied to the affected eye every one hour while awake for 1 week, then every 2 hours while awake until three weeks after enrollment.
  400 mg BID PO on study day one (loading dose), then 200 mg BID PO until 3 weeks from enrollment for patients weighing greater than 50 kg. For patients 40-50 kg, the loading dose is 300 mg BID PO on study day 1, then 150 mg BID PO until 3 weeks from enrollment. For patients weighing <40 kg, the loading dose is 200 mg BID PO, then 100 mg BID PO until 3 weeks after enrollment.
  Arms: Oral Voriconazole
Drug: Placebo — 1% voriconazole (topical) plus 0.01% preservative, 1 drop applied to the affected eye every one hour while awake for 1 week, then every 2 hours while awake until three weeks after enrollment.
  5% natamycin (topical), 1 drop applied to the affected eye every one hour while awake for 1 week, then every 2 hours while awake until three weeks after enrollment.
  Two tablets BID PO on study day one, then one tablet BID PO until 3 weeks from enrollment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the addition of oral voriconazole to topical treatment regimens results in lower rates of perforation in severe fungal corneal ulcers.

DETAILED DESCRIPTION:
Fungal corneal ulcers tend to have very poor outcomes with commonly used treatments. There has only been a single randomized trial of anti-fungal therapy for mycotic keratitis, and no new ocular anti-fungal medications have been approved by the FDA since the 1960s. The triazole voriconazole has recently become the treatment of choice for systemic fungal infections such as pulmonary aspergillosis. The use of topical ophthalmic preparations of voriconazole has been described in numerous case reports, however there has been no systematic attempt to determine whether it is more or less clinically effective than natamycin. Additionally, there have been many case reports of the use of oral voriconazole in the treatment of fungal corneal ulcers, however there has been no systematic attempt to determine if it improves outcomes in severe ulcers.

This study is a randomized, double-masked, placebo-controlled trial to determine if the use of oral voriconazole in severe ulcers reduces the rate of perforations. 240 fungal corneal ulcers with baseline visual acuity worse than 6/120 presenting to the Aravind Eye Hospitals and the UCSF Proctor Foundation will be randomized to receive oral voriconazole plus topical voriconazole and topical natamycin, or oral placebo plus topical voriconazole and topical natamycin. The primary outcome is the rate of perforation over the three month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a corneal ulcer at presentation
* Evidence of filamentous fungus on smear (KOH wet mount, Giemsa, or Gram stain)
* Visual acuity worse than 6/120 (20/400, logMAR 1.3)
* The patient must be able to verbalize a basic understanding of the study after it is explained to the patient, as determined by physician examiner. This understanding must include a commitment to return for follow-up visits.
* Willingness to be treated as an inpatient or to be treated as an outpatient and return every 3 days +/- 1 day until re-epithelialization and every week to receive fresh medication for 3 weeks
* Appropriate consent

Exclusion Criteria:

* Evidence of bacteria on Gram stain at the time of enrollment
* Evidence of acanthamoeba by stain
* Evidence of herpetic keratitis by history or exam
* Corneal scar not easily distinguishable from current ulcer
* Age less than 16 years (before 16th birthday)
* Bilateral ulcers
* Previous penetrating keratoplasty in the affected eye
* Pregnancy (by history or urine test) or breast feeding (by history)
* Known liver disease, including hepatitis or cirrhosis (Child-Pugh A-C)
* Acuity worse than 6/60 (2/200) in the fellow eye (note that any acuity, uncorrected, corrected, pinhole, or BSCVA 6/60 or better qualifies for enrollment)
* Acuity better than 6/120 (20/400) in the study eye (note that any acuity, uncorrected, corrected, pinhole, or BSCVA can be used for enrollment)
* Currently on rifampin, rifabutin, ritonavir, long acting barbiturates, phenytoin, carbamazepine, or other drugs known to interact with voriconazole
* Known allergy to study medications (antifungal or preservative)
* No light perception in the affected eye
* Not willing to participate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-05; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NV Prajna, DNB, FRC Ophth, Principal Investigator — Aravind Eye Hospitals; Nisha Acharya, MD, MS, Principal Investigator — Proctor Foundation, UCSF; Tom Lietman, MD, Principal Investigator — Proctor Foundation, UCSF
Locations (7):
- Proctor Foundation, UCSF, San Francisco, California, United States
- India (4):
  - Aravind Eye Hospital, Coimbatore, Tamil Nadu
  - Aravind Eye Hospitals, Madurai, Tamil Nadu
  - Aravind Eye Hospital, Pondicherry, Tamil Nadu
  - Aravind Eye Hospital, Tirunelveli, Tamil Nadu
- Nepal (2):
  - Bharatpur Eye Hospital, Bharatpur, Chitwan
  - Lumbini Eye Institute, Siddharthanagar, Lumbini

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zegans ME, Kamath MM, Jones JT, Bao R, Ross BS, Gutierrez-Perez C, Adams EM, Lightfoot JD, Poimenidou G, Pavuluri C, Prajna V, Cramer RA, Fuller KK. Propranolol is efficacious against Aspergillus and Fusarium corneal isolates in vitro and in a murine model of Aspergillus keratitis. Antimicrob Agents Chemother. 2025 Jun 4;69(6):e0166424. doi: 10.1128/aac.01664-24. Epub 2025 May 15. PMID 40372030

RESULTS

PARTICIPANT FLOW:
Period: 3-week Followup Visit
Arm/Group | Placebo | Oral Voriconazole
Started | 121 | 119
Completed | 112 | 113
Not Completed | 9 | 6
Not completed — Lost to Follow-up | 9 | 6
Period: 3-month Follow-up Visit
Arm/Group | Placebo | Oral Voriconazole
Started | 112 | 113
Completed | 100 | 107
Not Completed | 12 | 6
Not completed — Lost to Follow-up | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Oral Voriconazole | Total
Number analyzed (Participants) | 121 | 119 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 93 | 191
  >=65 years | 23 | 26 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [45 to 60] | 54 [42 to 62] | 54 [45 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 54 | 104
  Male | 71 | 65 | 136
Region of Enrollment [Number; unit: participants]
  Nepal | 98 | 98 | 196
  India | 23 | 21 | 44
Weight (lbs) [Median (Inter-Quartile Range); unit: lbs] | 108 [97 to 121] | 105 [94 to 123] | 108 [97 to 121]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Perforation or Therapeutic Penetrating Keratoplasty
Description: Hazard ratio of perforation or therapeutic penetrating keratoplasty (TPK) comparing voriconazole to placebo
Time Frame: 3 months from enrollment
Population: Comparison of rate of perforation or TPK between the treatment groups (topical voriconazole with oral voriconazole vs. topical voriconazole with oral placebo)
Measure: Number; unit: New perforations or TPK/person-days
Groups:
- Oral Voriconazole: oral voriconazole plus topical antifungal agents
- Oral Placebo: oral placebo plus topical antifungal agents
Arm/Group | Oral Voriconazole | Oral Placebo
Number analyzed (Participants) | 119 | 121
New perforations or TPK/person-days | 0.0095562 | 0.011204
Statistical Analysis 1: Comparison: Oral Voriconazole vs Oral Placebo; The sample size was determined based on the primary end point: perforation or the need for TPK within 3 months. Simulation-based analyses estimated that a sample sizeof 240 study participants (120 per arm) would provide 80% power to detect a 15% difference in the 3-month perforation or need for TPK rate between topical antifungal plus oral voriconazole vs topical antifungal alone,with a 2-tailed α value of .05 and approximately 15%loss to follow-up; Test type: Superiority; p = 0.29, Regression, Cox; Cox proportional hazards regression to estimate the hazard of perforation or need for TPK; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.57 to 1.18]

2. Secondary Outcome: Best Spectacle-corrected logMAR Visual Acuity
Description: Best spectacle-corrected logMAR visual acuity at 3 months after enrollment, adjusting for enrollment BSCVA and treatment arm in a multiple linear
Time Frame: 3 months after enrollment
Population: Best spectacle-corrected logMAR visual acuity at 3 weeks after enrollment, adjusting for enrollment BSCVA and study site
Measure: Mean (Standard Error); unit: logMAR
Arm/Group | Oral Voriconazole | Oral Placebo
Number analyzed (Participants) | 107 | 100
logMAR | .7852594 (.1083858) | .787141 (.1646131)

3. Secondary Outcome: Best Spectacle-corrected logMAR Visual Acuity at 3-weeks
Description: Best spectacle-corrected logMAR visual acuity at 3 weeks after enrollment, adjusting for enrollment BSCVA and treatment arm in a multiple linear
Time Frame: 3 weeks after enrollment
Population: as for outcome 2
Measure: Mean (Standard Error); unit: logMAR
Arm/Group | Oral Voriconazole | Oral Placebo
Number analyzed (Participants) | 113 | 112
logMAR | .8745454 (.1080198) | .744252 (.0964871)

4. Secondary Outcome: Size of Infiltrate/Scar - 3 Months
Description: Size of infiltrate/scar at 3 months after enrollment, using enrollment infiltrate scar/size as a covariate
Time Frame: 3 months after enrollment
Population: Mean infiltrate scar size at three months correcting for baseline scar size and site
Measure: Mean (Standard Error); unit: mm^2
Groups:
- Oral Voriconazole: Oral voriconazole treated participants
Arm/Group | Oral Voriconazole | Oral Placebo
Number analyzed (Participants) | 107 | 100
mm^2 | .9319315 (.06508) | .697005 (.0927)

5. Secondary Outcome: Size of Infiltrate/Scar
Description: Size of infiltrate/scar at 3 weeks after enrollment, using enrollment infiltrate scar/size as a covariate
Time Frame: 3 weeks after enrollment
Population: Mean infiltrate scar size at three weeks.
Measure: Mean (Standard Error); unit: mm^2
Groups:
- Oral Placebo: Oral Placebo plus topical antifungal agent
Arm/Group | Oral Voriconazole | Oral Placebo
Number analyzed (Participants) | 113 | 112
mm^2 | .2192398 (.1663) | .7973467 (.073885)

6. Secondary Outcome: Hazard Ratio for Re-epithelialization
Description: Hazard Ratio of re-epithelialization comparing the treatment groups
Time Frame: Up to 21 days
Measure: Number; unit: Number re-epthelialized/person-days
Groups:
- Oral Voriconazole: oral voriconazole plus topical antifungal
- Oral Placebo: oral placebo plus topical antifungal
Arm/Group | Oral Voriconazole | Oral Placebo
Number analyzed (Participants) | 113 | 112
Number re-epthelialized/person-days | .0141123 | .0130862
Statistical Analysis 1: Comparison: Oral Voriconazole vs Oral Placebo; Test type: Superiority; p = 0.65, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [.49 to 1.57]

7. Secondary Outcome: Microbiological Cure at 7 Days
Description: Fungal Culture negative at 7 days post treatment
Time Frame: 7 days
Population: Fungal Culture negative at 7 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Oral Voriconazole
Number analyzed (Participants) | 121 | 119
Participants | 50 | 50

8. Secondary Outcome: Number of Adverse Events
Description: Comparing the number of serious and non-serious adverse events by treatment arm.
Time Frame: 3-months from enrollment
Measure: Number; unit: adverse events
Arm/Group | Oral Voriconazole | Placebo
Number analyzed (Participants) | 119 | 121
adverse events | 58 | 28
Statistical Analysis 1: Comparison: Oral Voriconazole vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact — Statistically significant after Holms-Šidák correction for multiple comparisons

9. Secondary Outcome: Minimum Inhibitory Concentration of Isolates - Natamycin
Description: Minimum Inhibitory Concentration (MIC) of isolates to natamycin by treatment arm
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Oral Voriconazole | Placebo
Number analyzed (Participants) | 62 | 64
mg/L | 12 [4 to 32] | 4 [4 to 16]

10. Secondary Outcome: Minimum Inhibitory Concentration of Isolates - Voriconazole
Description: Minimum Inhibitory Concentration (MIC) of isolates to voriconazole by treatment arm
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Oral Voriconazole | Placebo
Number analyzed (Participants) | 62 | 64
mg/L | 1 [0.5 to 4] | 2 [0.5 to 4]

ADVERSE EVENTS:
Time Frame: Over the entire course of the trial. (June, 2010-December 2015)
Arm/Group | Placebo | Oral Voriconazole
Serious Adverse Events (participants affected / at risk) | 1/121 | 7/119
Other Adverse Events (participants affected / at risk) | 27/121 | 52/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | Oral Voriconazole (N=119)
Endophthalmitis (Eye disorders) | 1 | 3
Evisceration (Eye disorders) | 0 | 1
Myocardial infarction or stroke (Cardiac disorders) | 0 | 1
AST or ALT elevated to five times the upper limit of normal (Hepatobiliary disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=121) | Oral Voriconazole (N=119)
Ulcer not healing after 6 weeks of therapy (Eye disorders) | 2 | 5
Increase in hypopyon (increase>2mm) (Eye disorders) | 8 | 5
Headache (General disorders) | 8 | 7
AST or ALT elevated to twice upper limit of normal (Hepatobiliary disorders) | 0 | 8
Dizziness (General disorders) | 1 | 5
Vomiting (General disorders) | 2 | 4
Visual disturbances (Psychiatric disorders) | 0 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 3
Fever (General disorders) | 2 | 2
Lethargy (General disorders) | 1 | 2
Nausea (General disorders) | 1 | 2
Local allergic reaction (General disorders) | 1 | 1
Other systemic event thought to be related to study drug (General disorders) | 0 | 1
Dermatologic reaction (General disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No